CLINICAL TRIAL: NCT00384527
Title: Multicenter, Double-blind Study of Nitazoxanide Compared to Vancomycin in the Treatment of Clostridium Difficile-associated Disease
Brief Title: Study of Nitazoxanide in the Treatment of Clostridium Difficile-associated Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated early due to slow recruitment.
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Romark Laboratories, L.C., Romark Laboratories, L.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM01-3032
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2008-10

CONDITIONS: Clostridium Infections
Keywords: Clostridium difficile
MeSH Terms: conditions — Clostridium Infections | interventions — nitazoxanide; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Nitazoxanide
- 2 (Active Comparator)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Nitazoxanide — One nitazoxanide 500 mg tablet twice daily plus one vancomycin-placebo capsule four times daily for 10 days.
  Other Names: Alinia
  Arms: 1
Drug: Vancomycin — One vancomycin 125 mg capsule four times daily plus one nitazoxanide-placebo twice daily for 10 days.
  Other Names: VANCOCIN
  Arms: 2

SUMMARY:
The primary objective of the study is to demonstrate non-inferiority of nitazoxanide compared to vancomycin in resolving symptoms of Clostridium difficile-associated disease (CDAD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients with new onset of disease evidenced by diarrhea (≥ 3 unformed stools within 24 hours), and one or more of the following symptoms of CDAD:

  * abdominal pain or cramps
  * peripheral leukocytosis
  * fever
* C. difficile toxin A or B detected in a stool specimen obtained within 3 days before enrollment by enzyme immunoassay.
* Patients willing to avoid the following medications during the study:

  * oral and intravenous metronidazole
  * oral vancomycin
  * anti-peristaltic drugs
  * opiates (patients on opiates may be included in the study if they were taking opiates prior to enrollment and the dose is not increased during the study)
  * Saccharomyces cerevisiae (baker's yeast)
  * Lactobacillus GG
  * cholestyramine
  * colestipol

Exclusion Criteria:

* Patients with other known causes of diarrhea or colitis (e.g., Shigella, Salmonella, Cryptosporidium parvum, Giardia lamblia, Entamoeba histolytica, inflammatory bowel disease, irritable bowel syndrome, advanced AIDS or chemotherapy for malignancy).
* Patients that commonly have 3 or more stools per day and/or severe abdominal pain in the absence of CDAD.
* Patients with severe lactose intolerance.
* Patients with more than 1 recurrence of CDAD during the 6 months prior to enrollment.
* Patients unable to take oral medications.
* Use within 1 week of enrollment of any drug or therapy with anti-C. difficile activity such as oral or intravenous metronidazole and oral vancomycin. [Patients that have taken up to 3 doses of metronidazole or vancomycin can be included in the study].
* Females of child bearing age who are either pregnant, breast-feeding or not using birth control and are sexually active.
* Patients who are either clinically unstable (e.g., fulminant disease patients with signs of toxic megacolon, imminent perforation, colectomy or death) or unlikely to live throughout the 31-day duration of the study due to underlying illness.
* History of hypersensitivity to nitazoxanide or vancomycin or any active ingredient in the formulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinical response (resolution of all symptoms of CDAD) | End of treatment (day 12-14 after beginning treatment)

SECONDARY OUTCOMES:
Time from first dose to resolution of symptoms of CDAD | Any time after beginning treatment and must be sustained through end of treatment visit
Microbiological Recurrence | Clinical response at end of treatment visit with recurrence of symtpoms prior to study day 31 and C. difficile toxins detected in stool.
Sustained clinical response | End of treatment response sustained through study day 31.
Clinical Recurrence | Clinical response at the end of treatment with recurrent symptoms of CDAD prior to study day 31, but no C. difficile toxins detected.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Kauffman, MD, Principal Investigator — John D. Dingell VAMC; Adam Bressler, MD, Principal Investigator — Atlanta Institute for Medical Research; Wesley Bray, MD, Principal Investigator — Wellstar Clinical Trials; James Grendell, MD, Principal Investigator — Winthrop University Hospital; Bradley Allen, MD, Principal Investigator — Richard L. Roudebush VA Medical Center; Partha Nandi, MD, Principal Investigator — Center for Digestive Health; Daniel Musher, MD, Principal Investigator — Michael E. Debakey VAMC; Julia Garcia-Diaz, MD, Principal Investigator — Oschner Clinic Foundation; David Rand, MD, Principal Investigator — Torrence Memorial Hospital; David Johnson, MD, Principal Investigator — Bay Pines VAMC
Locations (10):
- United States (10):
  - Torrance Memorial Hospital, Torrance, California
  - Bay Pines VAMC, Bay Pines, Florida
  - Atlanta Institute for Medical Research, Atlanta, Georgia
  - Wellstar Clinical Trials, Atlanta, Georgia
  - Richard L. Roudebush VAMC, Indianapolis, Indiana
  - Oschner Clinic Foundation, New Orleans, Louisiana
  - John D. Dingell VAMC, Ann Arbor, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Winthrop University Hospital, Mineola, New York
  - Michael E. Debakey VAMC, Houston, Texas

REFERENCES:
- [Derived] Musher DM, Logan N, Bressler AM, Johnson DP, Rossignol JF. Nitazoxanide versus vancomycin in Clostridium difficile infection: a randomized, double-blind study. Clin Infect Dis. 2009 Feb 15;48(4):e41-6. doi: 10.1086/596552. PMID 19133801